CLINICAL TRIAL: NCT00342121
Title: Influence of Corn Farming on the Immune System
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902197; 02-C-N197
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: NHL
Keywords: Cancer; NHL; Pesticides; Atrazine; Organophosphates; Cancer Risk; Normal Control
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: Corn farmers enrolled in the Agricultural Health Study who are non-smokers, and who plan to apply specific pesticides.
- 2: Control subjects selected from agricultural extension workers in Iowa who are non-smokers

SUMMARY:
This study will look for links between corn farming practices and short-term changes in immune function in farmers throughout the growing season. It will examine biologic effects associated with specific pesticide exposures and general planting activities, such as tillage. Farmers have an increased risk of non-Hodgkin s lymphoma and certain other blood cancers such as multiple myeloma and leukemia, but the reasons for this increase have not been identified. Findings of this study may contribute to learning the causes of cancers such as non-Hodgkin s lymphoma.

Farmers enrolled in the Agricultural Health Study (a study of pesticide applicators and their spouses in Iowa and North Carolina) and a group of control subjects selected from agricultural extension workers in Iowa may participate in this study.

The study involves six home visits to farmers and four visits to farmers to individuals in the control group. All participants will complete the following tests and procedures:

* Questionnaires and diaries During the first visit, all participants will have a medical history review, including questions about smoking and other health habits. Farmers will be asked about their farming practices, and controls will be asked about their occupations. Farmers will fill out daily diaries during short time periods of interest around certain pesticide applications to describe farming activities that day. At other times during the growing season before harvest, farmers will fill out weekly diaries describing farming activities; controls, meanwhile, will fill out weekly diaries describing their health and work activities. At home visits during the farmers growing season, all participants will fill out questionnaires about their health. Finally, farmers and controls will complete a more extensive questionnaire in the off-season, during the last home visit, to learn about their activities and exposures in the final part of the year (post-harvest for farmers).
* Urine samples: At the time of each home visit, controls will provide a urine sample that the interviewer will take that day. Farmers, too, will provide urine samples at the time of home visits, but they will also collect urine samples for a period of 4 days each during short time periods of interest after certain pesticide applications. The interviewer will collect these samples immediately at the end of these periods.
* Blood samples: At the time of each home visit, the interviewer will draw 50 ml (3.5 tablespoons) of blood.
* Telephone calls: Farmers will be called frequently from once every 2 weeks to every other day to schedule visits at the times of interest. Control subjects will also be called frequently to schedule their visits closely to those of the farmers.

DETAILED DESCRIPTION:
When compared to the general population, farmers have an increased risk of non-Hodgkin's lymphoma (NHL) and certain other hematopoeitic cancers (i.e., multiple myeloma, leukemia). Factors that contribute to this excess risk have not been discerned. While several epidemiologic studies have observed an increased risk of NHL among farmers who are exposed to certain pesticides (i.e., phenoxyacetic acids, organophosphates, organochlorines, and triazines), these studies have not been conclusive. In addition, a clear mechanistic association between farming or pesticide exposure and subsequent development of cancer has not been identified. Given that immunocompromised individuals are at increased risk for NHL, it has been hypothesized that altered immune function may be an indicator of increased potential for the development of immunologically based diseases such as NHL. Therefore, research into early immunologic effects of farming exposures holds some promise in discerning disease mechanisms and in identifying specific etiologic agents for lymphatic cancers such as NHL. Few such studies have been conducted.

This protocol outlines a study of immune effects among corn farmers within Agricultural Health Study (AHS) cohort. The main objective is to evaluate the changes in immune parameters in farmers throughout the growing season, as well as effects of specific pesticide exposures including atrazine and organophosphate (OP) insecticides. Farmers and control subjects were contacted just prior to planting (February-March) to be enrolled in the study. Biological sampling before and after planting and application of preemergent pesticides (likely to include atrazine and possibly Ops or carbamates) allowed examination of short-term biologic effects associated with specific pesticide exposures and general planting activities (e.g., tillage). The first post-emergent application of organophosphate insecticide will also be monitored, in order to evaluate short-term biologic effects associated with this OP exposture. Post-harvest and off-season samples also were collected to allow evaluation of overall immune effects of farming activities. Pesticide exposures (e.g., atrazine, OPs, and potentially 2,4-D or carbamates) are being assessed primarily by measurement of the parent compound or its metabolites in urine, and additional information on farming activities and work practices will be obtained by questionnaire. Farmers serve as their own self-controls, and a selected control group will provide a means for external comparison.

ELIGIBILITY:
* INCLUSION CRITERIA:

Male corm farmers in the AHS who plan to apply specific pesticides.

Any ethnicity or race groups are included.

Limit the age criteria for inclusion to 40 to 60 years.

Only non-smokers are included in the study.

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Farmers enrolled in the Agricultural Health Study and a group of control subjects selected from agricultural extension workers in Iowa may participate in this study. Specifically, male corm farmers in the AHS who plan to apply specific pesticides. Only non-smokers are included in the study.@@@
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2002-05-03; Primary Completion 2004-01-31 (Actual); Study Completion 2008-02-05 (Actual)

PRIMARY OUTCOMES:
Immunilogical effects of farming exposues | Before and after application of pesticies
  Evaluate the changes in immune parameters in farmers throughout the growing season, as well as effects of specific pesticide exposures including atrazine and organophosphate (OP) insecticides. Pesticide exposures (e.g., atrazine, OPs, and potentially 2,4-D or carbamates) are being assessed primarily by measurement of the parent compound or its metabolites in urine, and additional information on farming activities and work practices will be obtained by questionnaire. Farmers serve as their own self-controls, and a selected control group will provide a means for external comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Beane-Freeman, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Iowa, Iowa City, Iowa, United States